CLINICAL TRIAL: NCT05993988
Title: The Effect of Telerehabilitation Practice on the Clinical Stress Level and Stress Responses of Nursing Students During Their First Clinical Experience
Brief Title: The Effect of Telerehabilitation on Clinical Stress Level and Stress Responses in Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Mustafa Savaş Torlak, Ass. Prof., KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Karatayanxiety
Record Dates: First submitted 2023-08-04; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Stress
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: parallel assignment
Who Masked: Participant
Masking Description: single
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): The participants in the control group did not receive any intervention.
- Exercise group (Experimental): The participants in the exercise group performed Jacobson muscle relaxation exercises with a specialist physiotherapist through the Zoom program (https://zoom.us). The exercises were applied 4 days a week for 4 weeks.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Muscle relaxing Technique
  Arms: Exercise group

SUMMARY:
It was aimed to examine the effect of telerehabilitation on clinical stress level and stress responses in nursing students.

DETAILED DESCRIPTION:
It was aimed to examine the effect of telerehabilitation on clinical stress level and stress responses in nursing students.There is no study in the literature examining the relationship between telerehabilitation and clinical stress in nursing students. Since our study will be the first to investigate the subject, we foresee that it is scientifically important and will shed light on future studies. In addition, national or international publications are planned after the study is completed.

ELIGIBILITY:
Inclusion Criteria:

* to be between the ages of 18-24
* to do the first clinical internship in the hospital

Exclusion Criteria:

* have joint limitation
* have congenital anomaly
* have any orthopedic problem
* have any serious psychological problems

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale for Nursing Students | baseline and 4 weeks
  Sheu et al. (2002) originally in Chinese, the scale consists of 29 items.Total score; It ranges from 0 to 116. A high score indicates a high level of stress. The internal consistency coefficient value of the original scale is 0.86.
Biopsychosocial Response Scale of Nursing Students | baseline and 4 weeks
  The scale was developed by Sheu et al. (2002). There are 21 items in the scale.Total score; It ranges from 0 to 84 (sub-dimension total scores are 32, 28, and 24 points, respectively). High score indicates more symptom presence and poor bio-psycho-social status.

CONTACTS AND LOCATIONS:
Locations (1):
- Mustafa Savaş Torlak, Karatay, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided